CLINICAL TRIAL: NCT06774677
Title: Decoding the Extracellular Vesicles-driven Communication in the Microenvironment of Hairy Cell Leukemia to Improve Patient Care Management
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: HCL-EV; PNRR-TR1-2023-12377450 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Hairy Cell Leukemia (HCL)
MeSH Terms: conditions — Leukemia, Hairy Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a national multi-centre, experimental, cross-sectional, non-profit study.

DETAILED DESCRIPTION:
Extracellular vesicles are small particles circulating in plasma and documented as key players of intercellular crosstalk thanks to their cargo of proteins, lipids, and nucleic acids. The driving hypothesis of this study is that in Hairy Cell Leukemia-derived extracellular vesicles contribute to the maintenance of the tumor clone through regulation of selected key cells of the tumor microenvironment including immune cells and stromal cells, likely favoring immune evasion and marrow fibrosis. As a consequence, these circulating particles may be instrumental at identifying a biology-related, disease-specific and extracellular vesicle-based signature associated to outcomes.

ELIGIBILITY:
Inclusion criteria for patients:

* WHO2022-defined diagnosis of Hairy Cell Leukemia.
* Age ≥18 years.
* Signed informed consent.

Inclusion criteria for Healthy Donors:

* Age ≥18 years.
* Volunteers in general good health, free from any disease or serious illness.
* Signed informed consent.

Exclusion criteria

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed by Hairy Cell Leukemia patients subdivided as newly diagnosed (n=10), relapsed meeting treatment indications (N=5) and in complete response >2 years (N=10) and by Healthy Donors (n=25), enrolled among volunteers through the non-profit organization AIL Bologna ODV.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Extracellular vesicle characterization | 1 years
  Verify whether hairy cell leukemia patients at different status (at diagnosis, in complete remission > 2 years, or relapsed meeting treatment indications) display specific extracellular vesicle-based signatures.

SECONDARY OUTCOMES:
Functional effects of extracellular vesicles | 1 years
  Elucidate whether plasma-derived extracellular vesicles of hairy cell leukemia patients and healthy donors and in vitro hairy cell-derived extracellular vesicles may functionally educate the immune microenvironment. Elucidate whether plasma-derived extracellular vesicles of patients and healthy donors may functionally affect the isolated hairy cells. Understand whether plasma-derived extracellular vesicles of patients and healthy donors and in vitro hairy cell-derived extracellular vesicles might shape the stromal microenvironment toward fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Catani, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo, PA
  - Policlinico Santa Maria alla Scotte, Siena, SI
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna